CLINICAL TRIAL: NCT02403791
Title: A Prospective, Multi-center, Open-label and Double-blind, Standard-controlled, Non-inferiority, Diagnostic Study of Lung Ultrasound for Management of Mechanical Ventilation in Neonatal Acute Respiratory Distress Syndrome
Brief Title: Point-of-Care Bedside Lung Ultrasound Examination Advanced Trial Protocol
Acronym: PoCBLUEPlus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The second affiliated hospital of Jinan University School of Medicine (Unknown); First Affiliated Hospital of Chengdu Medical College (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Women and Children Health Hospital of Jiangsu Province (Unknown); Affiliated Hospital of Sichuan Vocational College of Health and Rehabilitation (Unknown); First Affiliated Hospital of Jinan University (Other); Yangzhou University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); The Sichuan Second Hospital of Guangxi Medical University (Unknown); Guangzhou General Hospital (Other); Nankai University School of Medicine (Other); Guangdong Medical College (Other); Chongqing Medical University (Other); Tsinghua University (Other); Guiyang Medical University (Other); Shenzhen Institutes of Advanced Technology Chinese Academy of Science (Unknown); Jiamusi University (Unknown); The University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Hong Liu, MD, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PoC-BLUE-Plus One
Record Dates: First submitted 2015-03-22; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lung Ultrasound (Experimental): In infants allocated to this arm Lung ultrasound for detection of ARDS will be performed before chest radiography.
  Interventions: Device: Linear Ultrasonic Sounder
- Chest Radiography (Active Comparator): In infants allocated to this arm chest radiography will be performed for the detection of indirect signs of ARDS without ultrasound evaluation.
  Interventions: Device: Bedside X-ray Machine

INTERVENTIONS:
Device: Linear Ultrasonic Sounder — Lung ultrasound evaluation is performed after clinical assessment and before chest radiography
  Other Names: Bedside Ultrasonography System
  Arms: Lung Ultrasound
Device: Bedside X-ray Machine — Chest Radiography is performed after clinical evaluation without using ultrasound assessment.
  Other Names: Chest X-ray System
  Arms: Chest Radiography

SUMMARY:
The purpose of this study was to evaluate the availability and diagnostic accuracy of point-of-care bedside lung ultrasound examination in management of mechanical ventilation in neonatal acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Neonatal acute respiratory distress syndrome (ARDS) is a critical condition requiring dynamic evaluation and interventions. Point-of-care bedside lung ultrasound examination (PoC-BLUE) is a noninvasive, readily available imaging modality that can complement physical and clinical evaluation.

At any time, most neonates and infants with ARDS in medical intensive care units (ICUs) require mechanical ventilation, making it one of the most frequently used critical care technologies. However, difficulties with regard to the accurate diagnosis of ARDS before administration of mechanical ventilation, dynamic monitoring of treatment effects during administration of mechanical ventilation, and decision-making of timing in weaning from mechanical ventilation, are often encountered in the majority neonates and infants who require mechanical ventilation.

Hence, techniques that expedite and advance the knowledge of the administration of mechanical ventilation should have an important clinical significance in the diagnosis, treatment and prognosis of ARDS.

Preliminary researches have suggested that BLUE has a high diagnostic accuracy in patients with acute respiratory failure, and has the potential to quantify the rate and degree of diaphragm thinning during mechanical ventilation, which may be useful to predict extubation success or failure during either spontaneous breathing (SB) or pressure support (PS) trials.

Unfortunately, few studies focus on the availability of PoC-BLUE in management of mechanical ventilation in neonatal acute respiratory distress syndrome. Also, they call into question the possible association of the demographic and clinical confounders with the diagnostic accuracy of PoC-BLUE for diagnosis, monitoring and prognosis of ARDS in the whole process of mechanical ventilation.

Given that a considerable need for a timely and dynamic diagnosis of severe condition and therapy evaluation during mechanical ventilation has been triggered to integrate the currently available bulk of knowledge and information, the objective of this study is to investigate the availability and diagnostic accuracy of PoC-BLUE Plus protocol in management of mechanical ventilation in ARDS.

ELIGIBILITY:
Inclusion Criteria:

* All infants who present to the ICU with respiratory symptoms suspicious for ARDS, according to Pediatric Acute Respiratory Distress Syndrome: Consensus Recommendations From the Pediatric Acute Lung Injury Consensus Conference, which is proposed by The Pediatric Acute Lung Injury Consensus Conference Group.
* In whom the treating Collaborative Review Groups of Poc-BLUE-Plus protocol believe would benefit from diagnostic imaging.

Exclusion Criteria:

* Infants who arrive at the ICU with a previously performed chest radiography
* Unstable infants with life-threatening injuries who require ongoing resuscitation

Ages: 1 Day to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of Lung Ultrasound in Neonatal ARDS | Accuracy will be measured at the end of clinical evaluation in the ICU, an expected average of 4 days
  Accuracy of lung ultrasound and chest radiography will be measured using as gold standard the independent evaluation of the entire medical records by two expert emergency physicians blinded to the lung ultrasound results and radiographic reports (digitalized chest radiography images will be available).

SECONDARY OUTCOMES:
Accuracy of Lung Ultrasound in the Ventilator-Associated Pneumonia | Accuracy will be measured at the end of clinical evaluation in the ICU, an expected average of 4 days
  Accuracy of lung ultrasound and chest radiography will be measured using as gold standard the independent evaluation of the entire medical records by two expert emergency physicians blinded to the lung ultrasound results and radiographic reports (digitalized chest radiography images will be available).
Accuracy of Lung Ultrasound in the Weaning of Ventilatory Support | Accuracy will be measured at the end of clinical evaluation in the ICU, an expected average of 4 days
  Accuracy of lung ultrasound and chest radiography will be measured using as gold standard the independent evaluation of the entire medical records by two expert emergency physicians blinded to the lung ultrasound results and radiographic reports (digitalized chest radiography images will be available).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, MD, Study Director — The First Affiliated Hospital with Nanjing Medical University

REFERENCES:
- [Result] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Result] Muscedere J, Dodek P, Keenan S, Fowler R, Cook D, Heyland D; VAP Guidelines Committee and the Canadian Critical Care Trials Group. Comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia: diagnosis and treatment. J Crit Care. 2008 Mar;23(1):138-47. doi: 10.1016/j.jcrc.2007.12.008. PMID 18359431
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Result] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959